CLINICAL TRIAL: NCT07390825
Title: Evaluation of the Effects of Aquatic Therapy on Activities of Daily Living, Walking, Balance, Posture, Pain, and Depression in Parkinson's Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Duygu Yanıktaş, Assistant Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TABED 1-25-938
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Aquatherapy; Rehabilitation of Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study was designed as a single-blind trial, where participants were kept unaware of their group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Control Group (Home-based Exercise) (Experimental): Control Group (Home-based Exercise)
  Interventions: Other: home exercise
- Arm2: Experimental Group (Experimental): Experimental Group (Aquatherapy + Home-based Exercise)
  Interventions: Other: Aquatherapy

INTERVENTIONS:
Other: Aquatherapy — The specific aquatic exercise protocol for Group 2, conducted in a 120 cm deep therapy pool at 30-32°C, includes the following exercises:
  Gait and Mobility: Water walking (forward and backward) and side-stepping.
  Dynamic Balance: Forward and lateral lunges, and single-leg stance/balance drills.
  Lower Extremity Strengthening: Hip kicks performed at the pool wall (flexion, extension, and abduction) and standing knee raises.
  Upper Body and Coordination: Arm raises (multi-directional) and deep-water cycling movements.
  Home Exercise Component: In addition to aquatic sessions, patients will continue land-based exercises including posture correction, flexibility/stretching, balance-coordination training, and strengthening.
  Arms: Arm2: Experimental Group
Other: home exercise — Group 1 patients will be prescribed a home exercise program at least 5 days per week for a duration of 6 weeks
  Arms: Arm 1: Control Group (Home-based Exercise)

SUMMARY:
Parkinson's Disease (PD) is a progressive neurodegenerative disorder characterized by motor symptoms such as bradykinesia, tremors, and postural instability, as well as various non-motor symptoms. Conventional land-based rehabilitation is standard; however, aquatherapy-utilizing water's buoyancy, hydrostatic pressure, and viscosity-offers a promising alternative to improve balance and mobility while reducing fall risks. This study aims to evaluate the effects of aquatherapy on gait, balance, posture, freezing of gait, activities of daily living (ADL), pain, and depression in Turkish PD patients.

This is a prospective, single-blind, randomized controlled trial involving 42 patients at Ankara City Hospital. Participants will be divided into two groups:

* Group 1 (Control): Home-based exercise program (5 days/week for 6 weeks).
* Group 2 (Intervention): Home-based exercises plus supervised aquatherapy (3 sessions/week, 45 minutes each, in a 30-32°C pool).

The study utilizes high-tech objective measurements and validated scales:

* Gait & Posture: Zebris Gait Analysis (spatiotemporal parameters) and Diers Formetric 4D (topographical posture analysis).
* Balance: HUR-Smart Balance device and the Berg Balance Scale.
* Clinical Scales: PDQ-39 (quality of life), Freezing of Gait Questionnaire, Falls Efficacy Scale, MMSE (cognitive), Beck Depression Inventory, and VAS (pain).

This research is noteworthy as the first aquatherapy study among Turkish PD patients to utilize a large sample size and standardized aquatic exercise protocols. It seeks to provide a comprehensive analysis of both motor and non-motor improvements, potentially establishing aquatherapy as a superior adjunctive treatment for enhancing functional independence in Parkinson's patients.

Primary hypothesis or outcome measure : Parkinson's Disease Questionnaire-39 . PDQ-39 is a patient-reported outcome measure designed to evaluate the health-related quality of life in Parkinson's patients across eight specific domains, including mobility, activities of daily living, and emotional well-being.

DETAILED DESCRIPTION:
Abstract / Project Description Parkinson's Disease (PD) is a progressive neurodegenerative disorder characterized by the degeneration of dopamine-producing cells in the substantia nigra, ranking as the second most common neurodegenerative disease after Alzheimer's. The prevalence of the disease in Turkey is approximately 2/1000. The primary symptoms of Parkinson's disease include bradykinesia, resting tremor, rigidity, and postural instability. Posture, balance, and gait disturbances are significant findings that emerge during the course of the disease, causing severe disability. The gait pattern in PD varies across different stages and affects patients to varying degrees. Typically, a shortening of step length, patients walk slowly with small steps. In advanced stages, difficulty in initiating gait, freezing of gait, and postural instability are frequently developing symptoms. In addition to classic motor findings, non-motor symptoms such as urinary incontinence, sexual dysfunction, orthostatic hypotension, sleep disorders, depression, anxiety, and pain may also be observed.

The Modified Hoehn & Yahr Staging is a scale used to stage Parkinson's disease, with proven validity and reliability in Turkish. Developed by Hoehn and Yahr in 1967, this system allows both the patient and the clinician to easily define the severity of the disease and evaluate its progression across five stages. In the literature, Stages 1 and 2 are classified as "mild," Stage 3 as "moderate," and Stages 4 and 5 as "severe".

As conventional rehabilitation therapy, Parkinson's patients are frequently prescribed land-based gait and mobilization, posture, relaxation exercises, occupational therapy, and respiratory and swallowing exercises. Whether combined with other therapies or not, aquatherapy improves balance and functional mobility in PD patients compared to conventional rehabilitation. Aquatherapy, developed to improve balance, make walking more functional, and minimize strength imbalances between muscles, is considered a viable method for PD .

Aquatherapy is a rehabilitation method based on exercises performed in water using the physical properties of water . It is beneficial in the treatment of musculoskeletal, neurological, and cardiopulmonary diseases, among other conditions. The therapeutic safety margin of aquatherapy is quite broad . During treatment, the physical properties of water are utilized: hydrostatic pressure increases lymphatic and venous return in the extremities, contributing to the reduction of edema. Due to the buoyancy of water, patients move more comfortably; body weight is reduced by 90% with immersion up to the cervical region and by 60% up to the xiphoid process . Because of water's viscosity, resistance to movement is higher than in air, allowing movements to be performed at a constant speed. This resistance makes water an effective environment for strengthening. Additionally, heat can be retained or transferred through the thermodynamic effect of water . Aquatherapy is recognized as an effective adjunctive treatment in PD, particularly for improving motor symptoms . It reduces pressure on the joints, alleviates pain, provides support during movement, and reduces the risk of falling, thereby helping patients improve their balance skills .

In this study, the aquatherapy exercise program will be conducted in a therapy pool with a depth of 120 cm. Patients will be recommended to wear aquatic shoes to prevent slipping. Access to the pool will be provided via a lift. The water temperature will be maintained at 30-32°C. The aim of this study is to investigate the effects of aquatherapy on gait, balance, posture, freezing, activities of daily living (ADL), pain, and depression in Parkinson's patients.

3. Expected Benefits and Risks of the Research In this study investigating the efficacy of aquatherapy in PD, patients will be divided into two groups: the first group will receive only home-based exercises, while the second group will receive aquatherapy for 45 minutes three days a week in addition to the home exercise program. The objective is to evaluate the efficacy of aquatherapy on ADLs, gait, balance, posture, pain, and depression.

Expected contributions to the literature include:

* Being the first aquatherapy study conducted among Turkish patients diagnosed with Parkinson's.
* Evaluating balance, gait, posture, depression, and pain within the same study.
* Utilizing a larger sample size compared to existing studies in the literature.
* Standardizing aquatherapy exercises for Parkinson's patients. Potential risks include patient non-compliance with the treatment, sensitivity to pool chemicals, and the development of exercise intolerance.

  4. Type, Scope, and Design of the Planned Research This study is designed as a prospective, single-blind, randomized controlled trial. Patients diagnosed with Parkinson's who apply to the Ankara City Hospital Physical Medicine and Rehabilitation Hospital outpatient clinic and meet the inclusion criteria will be included. Informed consent will be obtained from participants. Clinical and demographic data will be recorded. The 42 patients included in the study will be divided into two groups using the single-blinded sealed envelope technique.
* Group 1: Will perform home exercises at least 5 days a week for 6 weeks.
* Group 2: Will perform the home exercise program 5 days a week, plus aquatherapy exercises 3 days a week for 6 weeks under the supervision of a physiotherapist.

Patients will be evaluated before and after treatment. Home exercises for Group 1 include posture, flexibility and stretching, balance-coordination, strengthening, and gait exercises. For Group 2, in addition to home exercises, a pool prescription including water walking, side-stepping, forward and lateral lunges, single-leg stance/balance, hip kicks at the pool wall, deep-water cycling, arm raises, and standing knee raises will be implemented.

The following scales, which have proven Turkish validity and reliability, will be utilized in the study: Parkinson's Disease Questionnaire-39 (PDQ-39), Berg Balance Scale, Freezing of Gait Questionnaire, Falls Efficacy Scale, Mini-Mental State Examination (MMSE), Beck Depression Inventory, and the Visual Analog Scale (VAS), MDS-Unified Parkinson's Disease Rating Scale .

* Gait Analysis: Patients' gait patterns will be evaluated using the Zebris gait analysis system. Parameters to be measured include step length (distance between two consecutive footprints), step time (duration to complete a gait cycle), step width (mediolateral distance between ankle joint centers), walking speed, and cadence.
* Posture Analysis: Postural assessments will be conducted using the Diers Formetric 4D system, allowing for a comprehensive topographical analysis of the spine and pelvis.
* Balance Testing: Balance assessments will be performed using the HUR-Smart Balance device to provide objective data on stability and weight distribution.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Idiopathic Parkinson's Disease between the ages of 40-80 and consenting to the treatment.
* Being regularly followed by a neurologist and having a stable medical treatment regimen for at least 3 months.
* Having a disease stage between 1-3 according to the Modified Hoehn-Yahr Staging Scale (MHY).
* A score of 24 or higher on the Mini-Mental State Examination (MMSE).
* Being able to verticalize independently and ambulate with or without assistance.

Exclusion Criteria:

* Having orthopedic, rheumatological, or non-Parkinson's neurological disorders that affect functional status.
* Having a medical treatment regimen that has been modified within the last 3 months.
* Presence of Atypical Parkinson's Disease.
* Visual impairment.
* Presence of dementia.
* Decompensated cardiac or respiratory failure.
* Diabetes insipidus.
* Presence of systemic infection.
* Impaired skin integrity or the presence of skin infections.
* Increased sensitivity to inhaled steam or water chemicals.
* History of epilepsy or asthma.
* Urinary or fecal incontinence.
* Refusal to participate in or consent to the treatment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire-39 | From enrollment to the end of treatment at 6 weeks
  Patients' quality of life will be evaluated using the Parkinson's Disease Questionnaire-39 (PDQ-39).The PDQ-39 is a 39-item questionnaire that covers eight distinct dimensions of functioning and well-being. The domains include: Mobility , Activities of Daily Living, Emotional Well-being , Stigma, Social Support, Cognition, Communicatio, Bodily Discomfort.The questionnaire uses a 5-point Likert response format where patients rate their experiences from "never" (0) to "always" (4). For each of the eight dimensions, a score is calculated and normalized to a 0-100 scale using the formula:Dimension Score = (Sum of Item Scores / Maximum Possible Score for Dimension) × 100 each dimension the minimum possible score is 0 and the maximum possible score is 100 after normalization. Considering the entire PDQ-39, the raw total score ranges from 0 to 156, where 0 represents the best possible quality of life and 156 the worst possible quality of life.

SECONDARY OUTCOMES:
Berg Balance Scale | From enrollment to the end of treatment at 6 weeks.
  The Berg Balance Scale will be utilized to measure the patients' balance; the minimum possible total score on the Berg Balance Scale is 0, and the maximum possible score is 56. Higher scores indicate better balance performance, with 0 reflecting severe balance impairment and 56 representing normal balance function.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Uçan, Prof. Doctor, Study Director — Bilkent City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Bilkent City Hospital, Çankaya, Ankara
  - Bilkent City Hospital, Ankara, ÇANKAYA

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly to protect patient confidentiality and ensure strict adherence to personal data protection laws. The raw data contains sensitive health information that could potentially lead to the de-identification of participants, which would violate the ethical terms outlined in the informed consent forms

REFERENCES:
- [Background] Pinto C., et al. (2019). "The Effects of Hydrotherapy on Balance, Functional Mobility, Motor Status, and Quality of Life in Patients with Parkinson Disease: A Systematic Review and Meta-analysis", PM R, 11(3), 278-291. https://doi.org/10.1016/j.pmrj.2018.09.031
- See also: Exercise program is based on clinical guidelines provided by ChoosePT.com, the official consumer information website of the American Physical Therapy Association (APTA). — https://www.choosept.com/health-tips/10-exercises-in-pool